CLINICAL TRIAL: NCT03057652
Title: Algorithmic-Based Evaluation and Treatment Approach for Robotic Gait Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shuo-Hsiu Chang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0923
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Complete Spinal Cord Injury; Incomplete Spinal Cord Injury; Acquired Brain Injury; Multiple Sclerosis
MeSH Terms: conditions — Brain Injuries; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Each of the participants will receive training with each of the 3 wearable robotic exoskeletons (WRE) examined in this study, and the order of receipt will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- ReWalk, then EKSO, then REX (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX
- ReWalk, then REX, then EKSO (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX
- EKSO, then ReWalk, then REX (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX
- EKSO, then REX, then ReWalk (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX
- REX, then EKSO, then ReWalk (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX
- REX, then ReWalk, then EKSO (Experimental): Subjects will be asked to complete a screening visit, baseline and post assessment for each intervention training (ReWalk, EKSO, REX) and up to 15 training sessions per device.
  Interventions: Device: ReWalk; Device: EKSO; Device: REX

INTERVENTIONS:
Device: ReWalk — ReWalk is a type of wearable robotic exoskeleton (WRE). Subjects will be randomly assigned the order of participation in the exoskeleton devices.
  ReWalk training sessions will be scheduled for one hour to include don/doff of device, sit to stand, standing balance and walking. ReWalk phase will require 2 hours pre and 2 hours post training for outcome measurement assessments, plus a minimum of 5 training sessions, with the possibility of up to 15 training sessions to reach a minimal assistance level. The total time commitment for each subject will range from 14-20 weeks and cover 27-72 hours.
Device: EKSO — EKSO is a type of wearable robotic exoskeleton (WRE). Subjects will be randomly assigned the order of participation in the exoskeleton devices.
  EKSO training sessions will be scheduled for one hour to include don/doff of device, sit to stand, standing balance and walking. EKSO phase will require 2 hours pre and 2 hours post training for outcome measurement assessments, plus a minimum of 5 training sessions, with the possibility of up to 15 training sessions to reach a minimal assistance level. The total time commitment for each subject will range from 14-20 weeks and cover 27-72 hours.
Device: REX — REX is a type of wearable robotic exoskeleton (WRE). Subjects will be randomly assigned the order of participation in the exoskeleton devices.
  REX training sessions will be scheduled for one hour to include don/doff of device, sit to stand, standing balance and walking. REX phase will require 2 hours pre and 2 hours post training for outcome measurement assessments, plus a minimum of 5 training sessions, with the possibility of up to 15 training sessions to reach a minimal assistance level. The total time commitment for each subject will range from 14-20 weeks and cover 27-72 hours.

SUMMARY:
The purpose of this study is to develop an algorithmic-based evaluation and treatment approach for wearable robotic exoskeleton (WRE) gait training for patients with neurological conditions.

ELIGIBILITY:
Spinal Cord Injury Inclusion Criteria:

* Male or non-pregnant female
* ≥18 years of age
* Chronic (> 6 mo post) injury
* Diagnosis of spinal cord injury
* Able to achieve adequate fit within exoskeleton
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Weight <220 pounds
* Intact skin on all surfaces in contact with device and load bearing surfaces
* Ability to perform informed consent
* Cognitively intact and able to follow directions and demonstrate learning capability

Spinal Cord Injury Exclusion Criteria:

* Pregnancy
* Spinal instability
* Non-English speaking
* Unhealed limb or pelvic fractures or any condition restricting weight bearing in limbs
* Diagnosis of other neurological injury other than SCI such as CVA, MS, ABI, CP
* Uncontrolled spasticity (≥3 on Modified Ashworth Scale)[21]
* Colostomy
* Decreased range of motion or contractures in legs (>10° at hips, knees or ankles)
* Uncontrolled autonomic dysreflexia
* Unresolved deep vein thrombosis
* Inability to tolerate standing due to cardiovascular issues or orthostatic hypotension
* Severe comorbidities: active infections, heart, lung, or circulatory conditions
* Pressure sores, impaired skin integrity

Acquired Brain Injury(ABI) Inclusion Criteria:

* Male or non-pregnant female
* ≥18 years of age
* Chronic (> 6 mo post) injury
* Able to achieve adequate fit within exoskeleton
* Ability to perform informed consent
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Weight <220 pounds
* Intact skin on all surfaces in contact with device and load bearing surfaces
* Cognitively intact and able to follow directions and demonstrate learning capability

Acquired Brain Injury(ABI) Exclusion Criteria:

* Pregnancy
* Spinal instability
* Non-English speaking
* Unhealed limb or pelvic fractures or any condition restricting weight bearing in limbs
* Diagnosis of other neurological injury other than ABI such as SCI, MS, TBI, CP
* Decreased range of motion or contractures in legs (>10° at hips, knees or ankles)
* Inability to tolerate standing due to cardiovascular issues or orthostatic hypotension
* Pressure sores, impaired skin integrity
* Uncontrolled spasticity (≥3 on Modified Ashworth Scale)
* Colostomy
* Severe comorbidities: active infections, heart, lung, or circulatory conditions
* Unresolved deep vein thrombosis

Multiple Sclerosis (MS) Inclusion Criteria:

* Male or non-pregnant female
* ≥18 years of age
* Chronic (> 6 mo post) injury
* Diagnosis of multiple sclerosis
* Ability to perform informed consent
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Weight <220 pounds
* Able to achieve adequate fit within exoskeleton
* Intact skin on all surfaces in contact with device and load bearing surfaces
* Cognitively intact and able to follow directions and demonstrate learning capability

Multiple Sclerosis (MS) Exclusion Criteria:

* Pregnancy
* Spinal instability
* Non-English speaking
* Unhealed limb or pelvic fractures or any condition restricting weight bearing in limbs
* Decreased range of motion or contractures in legs (>10° at hips, knees or ankles)
* Inability to tolerate standing due to cardiovascular issues or orthostatic hypotension
* Uncontrolled autonomic dysreflexia
* Unresolved deep vein thrombosis
* Pressure sores, impaired skin integrity
* Uncontrolled spasticity (≥3 on Modified Ashworth Scale)
* Colostomy
* Severe comorbidities: active infections, heart, lung, or circulatory conditions[23,24]
* Diagnosis of other neurological injury other than MS such as CVA, SCI, ABI, CP
* MS Relapse in 3 months prior to recruitment

Able Bodied Inclusion Criteria:

* Male or non-pregnant female
* ≥18 years of age
* Weight <220 pounds
* Cognitively intact and able to follow directions and demonstrate learning capability[23]
* Healthy individuals with no history or diagnosis of neurological injury
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Able to achieve adequate fit within exoskeleton
* Intact skin on all surfaces in contact with device and load bearing surfaces
* Ability to perform informed consent[24]

Able Bodied Exclusion Criteria:

* Pregnancy
* Spinal instability
* Non-English speaking
* Unhealed limb or pelvic fractures or any condition restricting weight bearing in limbs
* Diagnosis of neurological injury such as CVA, SCI, ABI, CP, MS
* Decreased range of motion or contractures in legs (>10° at hips, knees or ankles)
* Severe comorbidities: active infections, heart, lung, or circulatory conditions
* Colostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in over ground gait speed as assessed by the 10 Meter Walk Test without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  The 10 Meter Walk Test (10MWT) will assess subject's self-selected gait speed.
Change in walking endurance as assessed by the 6 Minute Walk Test without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  The 6 Minute Walk Test (6MWT) assesses the distance walked in 6 minutes.
Change in muscle activity as assessed by electromyography (EMG) during 10MWT without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Surface EMG sensors will be placed on the skin of subjects' lower extremities during 10MWT.
Change in muscle activity as assessed by electromyography (EMG) during 6MWT without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Surface EMG sensors will be placed on the skin of subjects' lower extremities during 6MWT.
Change in energy expenditure as assessed by oxygen consumption during 10MWT without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Oxygen consumption will be calculated on a breath-by-breath basis measured by a portable metabolic system (Cosmed K4b2). This task will be performed during the 10MWT.
Change in energy expenditure as assessed by oxygen consumption during 6MWT without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Oxygen consumption will be calculated on a breath-by-breath basis measured by a portable metabolic system (Cosmed K4b2). This task will be performed during the 6MWT.
Change in gait kinematics as assessed by lower extremity joint excursion without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using motion capture system.
Change in gait kinematics as assessed by lower extremity joint angular velocities without WRE | within one week before start of WRE training, within 2 weeks after start of WRE training
  Infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using motion capture system.

SECONDARY OUTCOMES:
Bone mineral density as assessed by whole body scan | within one month before start of WRE training
  Subjects will undergo whole body bone scan according to standardized protocols.
Cognitive impairment as assessed by Folstein Mini Mental State Examination | within one month before start of WRE training
  Folstein Mini Mental State Examination provides information about orientation, attention, learning, calculation, delayed recall, and construction.
Lower Extremity Muscle Strength as assessed by using a force gauge such as a handheld dynamometer | within one month before start of WRE training
  We will measure lower extremity muscle strength using a force gauge such as a handheld dynamometer.
Spasticity as assessed by the Modified Ashworth Scale (MAS) | within one month before start of WRE training
  The Modified Ashworth Scale will be used to measure spasticity in lower limb.
Range of motion for lower extremity joints as assessed by manual examination | within one month before start of WRE training
  Range of joint motion of bilateral hip, knee and ankle joints. Subject will lie down on an examination table.
Stability during the maximum distance an individual can reach forward from a seated position as assessed by Modified Functional Reach (MFR) | within one month before start of WRE training
  Assesses a patient's stability by measuring the maximum distance an individual can reach forward from a seated position.
Walking ability in ambulatory individuals with SC as assessed by Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI): | within one month before start of WRE training
  Assesses functional walking ability in ambulatory individuals with SCI.
Amount of physical assistance needed for walking following paralysis resulted from SCI as assessed by Walking Index of Spinal Cord Injury (WISCI-II) | within one month before start of WRE training
  This test is performed by SCI population.
Motor recovery after stroke as assessed by Fugl-Meyer Assessment | within one month before start of WRE training
  Evaluates and measures recovery in post-stroke hemiplegic individuals.
Confidence in performing various ambulatory activities as assessed by Activities-Specific Balance Confidence Scale | within one month before start of WRE training
  Measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness. This is performed in ABI and MS population.
User feedback as assessed by a questionnaire | within one month before start of WRE training
  A questionnaire will be administered to allow participants to provide feedback regarding their experiences during intervention.
Over ground gait speed as assessed by the 10 Meter Walk Test while wearing WRE | within one month before start of WRE training
  The 10 Meter Walk Test (10MWT) will assess subject's self-selected gait speed. After WRE training has been completed, subjects will perform 10MWT while ambulating in the WRE.
Change in walking endurance as assessed by the 6 Minute Walk Test while wearing WRE | within one month before start of WRE training
  The 6 Minute Walk Test (6MWT) assesses the distance walked in 6 minutes. After WRE training has been completed, subjects will perform 6MWT while ambulating in the WRE.
Change in muscle activity as assessed by electromyography (EMG) during 10MWT while wearing WRE | within one month before start of WRE training
  Surface EMG sensors will be placed on the skin of subjects' lower extremities during 10MWT. After WRE training has been completed, subjects will be assessed by EMG during the 10MWT while ambulating in the WRE.
Change in muscle activity as assessed by electromyography (EMG) during 6MWT while wearing WRE | within one month before start of WRE training
  Surface EMG sensors will be placed on the skin of subjects' lower extremities during 6MWT. After WRE training has been completed, subjects will be assessed by EMG during the 6MWT while ambulating in the WRE.
Change in energy expenditure as assessed by oxygen consumption during 10MWT while wearing WRE | within one month before start of WRE training
  Oxygen consumption will be calculated on a breath-by-breath basis measured by a portable metabolic system (Cosmed K4b2). This task will be performed during the 10MWT. After WRE training has been completed, oxygen consumption will be assessed in subjects during the 10MWT while ambulating in the WRE.
Change in energy expenditure as assessed by oxygen consumption during 6MWT while wearing WRE | within one month before start of WRE training
  Oxygen consumption will be calculated on a breath-by-breath basis measured by a portable metabolic system (Cosmed K4b2). This task will be performed during the 6MWT. After WRE training has been completed, oxygen consumption will be assessed in subjects during the 10MWT while ambulating in the WRE.
Change in gait kinematics as assessed by lower extremity joint excursion while wearing WRE | within one month before start of WRE training
  Infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using motion capture system. After WRE training has been completed, subjects will be assessed while ambulating in the WRE.
Change in gait kinematics as assessed by lower extremity joint angular velocities while wearing WRE | within one month before start of WRE training
  Infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using motion capture system. After WRE training has been completed, subjects will be assessed while ambulating in the WRE.
Change in H-reflex of soleus muscle as assessed by electromyography (EMG) | within one week before start of WRE training, within 2 weeks after start of WRE training
  The tibialis nerve will be stimulated, and the size of each H-reflex will be measured as the peak-to-peak amplitude of the non-rectified EMG trace.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo-Hsiu Chang, PT, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States

REFERENCES:
- [Derived] Zhu F, Kern M, Fowkes E, Afzal T, Contreras-Vidal JL, Francisco GE, Chang SH. Effects of an exoskeleton-assisted gait training on post-stroke lower-limb muscle coordination. J Neural Eng. 2021 Jun 4;18(4). doi: 10.1088/1741-2552/abf0d5. PMID 33752175